CLINICAL TRIAL: NCT03466775
Title: Anti-Angiotensin II Type 1 Receptor Antibodies and Kidney Transplant Outcomes
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Collaborators: Center for Cardiovascular Research Berlin (Other)
Responsible Party: Principal Investigator, Carmen Lefaucheur, Professor, Paris Translational Research Center for Organ Transplantation
Other Study IDs: AT1R001
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: Kidney transplantation; Allograft rejection; Allograft survival; Anti-angiotensin II type 1 receptor antibody
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anti-angiotensin II type 1 receptor antibody measurement — Anti-angiotensin II type 1 receptor antibodies are assessed using quantitative ELISA in stored serum samples obtained within the first year after transplantation
Diagnostic Test: Measurement of ENDAT expression level allograft — Endothelial-associated transcript expression level is assessed using microarray in stored kidney allograft biopsies obtained within the first year after transplantation
Other: Allograft survival
Other: Allograft rejection appearance

SUMMARY:
Incompatibility between non-genetically identical donors and recipients has been increasingly recognized as the main contributing factor to solid allograft rejection and failure, through the triggering of donor-specific responses mediated by T- and B-lymphocytes. The Human Leucocyte Antigen (HLA) system has been identified as the main target of donor-specific responses, especially through the production by the recipient of antibodies directed toward non-self donor HLA molecules expressed on the allograft endothelium. As a consequence, in organ transplantation, the current approach to immunological risk stratification, patient monitoring and rejection diagnosis is based on biomarkers derived from the HLA system. However, this approach does not provide a sufficient accuracy for the risk stratification and the diagnosis of immunological complications in solid organ transplantation, which still remain the dominant cause of allograft failure.

A recent body of evidence supports that specific non-HLA antigens expressed on the allograft endothelium may be relevant to allograft rejection, suggesting that a new strategy to transplant diagnostic testing at a non-HLA level would help to overcome the limitations of the current HLA-based approach to immunological assessment of transplant recipients. Among antibodies to non-HLA endothelial antigens, angiotensin II type 1 receptor activating antibodies have been the most widely reported antibodies to associate with the occurrence of allograft rejection, dysfunction and loss, even if their independent role, with respect to the presence of concomitant anti-HLA antibodies, has not been demonstrated.

DETAILED DESCRIPTION:
The aims of this study are:

1. To assess the incidence of post-transplant anti-angiotensin II type 1 receptor antibodies within the first year after transplantation in an unselected population of kidney transplant recipients.
2. To investigate the incidence of biopsy-proven kidney allograft rejection according to the presence of post-transplant anti-angiotensin II type 1 receptor antibodies and of post-transplant concomitant donor-specific anti-HLA antibodies within the first year after transplantation, and to evaluate the incidence of rejection cases associated with anti-angiotensin II type 1-receptor antibodies that are not recognized by the current diagnostic approach based on HLA testing.
3. To investigate the allograft injury phenotype associated with post-transplant anti-angiotensin II type 1 receptor, using histopathology, immunochemistry and measurement of endothelial-associated transcript (ENDAT) expression level in allograft.
4. To evaluate the impact of post-transplant anti-angiotensin II type 1 receptor antibodies on kidney allograft survival up to 7 years after inclusion, in univariate and multivariable survival models including clinical, histological and immunological risk factors for allograft loss.

This study includes kidney recipients transplanted between January 1, 2008 and December 31, 2012 at Necker and Saint-Louis Hospitals (Paris, France), who undergo screening for post-transplant anti-angiotensin II type 1 receptor antibodies and simultaneous kidney allograft biopsy within the first year after transplantation, either at the time of an episode of rejection in the first year after transplantation or at 1 year after transplantation in the absence of previous rejection episode.

ELIGIBILITY:
Inclusion Criteria:

* Kidney recipient transplanted between January 1, 2008 and December 31, 2012
* Kidney recipient over 18 years of age
* Simultaneous histological and serological assessment within the first year after transplantation, including i) kidney allograft biopsy, ii) assessment of donor-specific anti-HLA antibodies, and available stored serum for anti-angiotensin II type 1 receptor antibody assessment

Exclusion Criteria:

* No simultaneous histological and serological assessment within the first year after transplantation, including i) absence of serum available for anti-angiotensin II type 1 receptor antibody assessment, and/or ii) absence of donor-specific anti-HLA antibody testing, and/or iii) absence of kidney allograft biopsy
* Inadequate kidney allograft biopsy according to the Banff classification for allograft rejection
* Combined transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes kidney recipients undergoing transplantation between January 1, 2008 and December 31, 2012 at Necker and Saint-Louis Hospitals (Paris, France).
Sampling Method: Non-Probability Sample
Enrollment: 1845 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-proven kidney allograft rejection according to the presence of post-transplant circulating anti-angiotensin II type 1 receptor antibodies within the first year after transplantation | One year after transplantation
  Anti-angiotensin II type 1 receptor antibody positivity is defined by serum concentration >10 U/mL using quantitative ELISA. Stratified analysis is performed according to the presence of post-transplant concomitant circulating donor-specific anti-HLA antibodies detected by single antigen bead assay in serum. Allograft rejection is defined on the basis of the 2015 update of the Banff classification for allograft rejection.
Comparison of allograft injury phenotype according to post-transplant anti-angiotensin II type 1 receptor antibody status and concomitant donor-specific anti-HLA antibody status | One year after transplantation
  Injury phenotype is based on histological allograft elementary lesions defined by the Banff classification (glomerulitis, peritubular capillaritis, interstitial inflammation, tubulitis, endarteritis, chronic allograft glomerulopathy, interstitial fibrosis, tubular atrophy, arteriosclerosis, arteriolar hyalinosis, C4d deposition in peritubular capillaries).
Association between the presence of post-transplant circulating anti-angiotensin II type 1 receptor antibodies and time to kidney allograft | Up to seven years after inclusion
  Univariate and multivariable models are performed, including adjustment for recipient age and gender, biopsy indication, glomerular filtration rate, proteinuria, presence of post-transplant circulating donor-specific anti-HLA antibodies and histological elementary lesions defined by the Banff classification, assessed at the time of antibody detection.

SECONDARY OUTCOMES:
Incidence of anti-angiotensin II Type 1 receptor antibodies in kidney transplant recipients within the first year after transplantation | One year after transplantation
  Anti-angiotensin II type 1 receptor antibody positivity is defined by serum concentration >10 U/mL using quantitative ELISA.
Comparison of endothelial-associated transcript expression (ENDAT) levels according to anti-angiotensin II type 1 receptor antibody status and donor-specific anti-HLA antibody status | One year after transplantation
  ENDAT expression levels are measured in kidney allograft biopsies performed at the time of antibody detection, showing microcirculation inflammation (sum of glomerulitis and peritubular capillaritis Banff scores >1), using microarray technology.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Lefaucheur, Principal Investigator — Paris Translational Research Center for Organ Transplantation; Alexandre Loupy, Principal Investigator — Paris Translational Research Center for Organ Transplantation; Duska Dragun, Principal Investigator — Clinic for Nephrology and Critical Care Medicine, Campus Virchow-Klinikum and Center for Cardiovascular Research, Medical Faculty of the Charité Berlin
Locations (2):
- France (2):
  - Kidney Transplant Department, Saint-Louis Hospital, Assistance Publique - Hôpitaux de Paris, Paris, France, Paris
  - Kidney Transplant Department, Necker Hospital, Assistance Publique - Hôpitaux de Paris, Paris, France, Paris

IPD SHARING:
Plan to Share IPD: No